CLINICAL TRIAL: NCT04745845
Title: The Impact of Noradrenaline on Ventriculo-arterial Coupling and Central Cardiovascular Energy Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019/287
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Heart Diseases
Keywords: Noradrenaline; Heart surgery; Intensive care; Cardiac physiology
MeSH Terms: conditions — Heart Diseases | interventions — Supine Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Noradrenalin (Experimental): treatment with 2 different NA concentrations in 2 different states of fluid responsiveness
  Interventions: Procedure: Noradrenalin

INTERVENTIONS:
Procedure: Noradrenalin — Norepinephrine challenge (concentration 'A' ) in fluid responsive position
  Other Names: Anti-Trendelenburg position/Semiupright position (20degr)
Procedure: Noradrenalin — Norepinephrine challenge (concentration 'A') in non-fluid responsive position
  Other Names: supine position
Procedure: Noradrenalin — Norepinephrine challenge (concentration 'B') in fluid responsive position
  Other Names: Anti-Trendelenburg position/Semiupright position (20degr)
Procedure: Noradrenalin — Norepinephrine challenge (concentration 'B') in non-fluid responsive position
  Other Names: supine position

SUMMARY:
The study aims to examine how noradrenaline in combination with venous return influences the energy transmission from heart to central circulation and arteries - also called arterio-ventricular coupling.

DETAILED DESCRIPTION:
After being informed about the study 40 elective CABG patients with written informed consent will undergo assessment of their arterio-ventricular coupling postoperatively after coronary bypass graft surgery. Whilst still in deep general anesthesia on the CT ICU the study population will be assessed by echocardiographic examination (transthoracic and transesophageal), blood pressure tracing by arterial line, respiratory data and ECG in 4 different situations.

Initially the individual patient is either considered fluid responsive (SVV >13%) og non- responsive (SVV<13%) by using stroke volume variation assessed by echocardiography.

In case of fluid responsiveness a fluid bolus of 4ml/kg of crystalloid fluid is given until SVV drops below 13% and the patient can be considered as fluid NON responder.

Right afterwards the study patient is stabilized with a baseline dose of noradrenaline (NA) intravenously in a supine position (situation 1). Situation 2 will be a slight increase in NA dose stabilizing mean arterial pressure in a "baseline + 20mmHg" state. After reversing the NA dose back to base line level the patient is allowed a short period of rest to wean of drug effect (4-5 x t1/2, appr. 12min). Subsequently the patient is to be placed in a 20% semi upright position (Anti-Trendelenburg) causing an increase in fluid responsiveness (situation 3). Following a phase of equilibration the dose of NA is again titrated up to obtain a 20mmHg increase in mean arterial pressure (situation 4).

There will be logging of arterial pressure curve and VTI-tracing I LVOT simultaneously (ultrapower, uPWR) as well as calculation of energy delivery, cardiac power, oscillatory power and -fraction and both arterial and ventricular elastance in every of those 4 situations.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary artery bypass graft surgery
* requirement for Noradrenaline/Norepinephrine

Exclusion Criteria:

* lack of informed consent
* patient unsuitable for mean arterial pressure (MAP) elevation of 20mmHg
* patient requiring different blood pressure range due to medical/surgical needs
* poor image quality due to patient factors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac Power | within 30 minutes after having been stabilised on the cardiothoracic ICU after performed CABG surgery
  Change in Cardiac Power in reaction to both different noradrenaline doses and states of fluid responsiveness.
  By logging invasive BP curve and tracing left ventricular outflow tract Velocity Time Integral (by echocardiography) simultaneously Total and Mean Cardiac Power (Watt) can be determined. Examining the response to different NA doses relative to fluid responsiveness the effect of NA on arterio-ventricular coupling can be examined.
Change in Oscillatory Power Fraction | within 30 minutes after having been stabilised on the cardiothoracic ICU after performed CABG surgery
  Change in Oscillatory Power Fraction (OPF) in reaction to both different noradrenaline doses and states of fluid responsiveness.
  By logging invasive BP curve and tracing left ventricular outflow tract Velocity Time Integral (by echocardiography) simultaneously Total Cardiac Power (TCP, Watt) and Cardiac Power Output (CPO, Watt) can be determined. By subtracting CPO from TCP, OPF (in %) can be calculated. Examining the response to different NA doses relative to fluid responsiveness the effect of NA on arterio-ventricular coupling can be examined.

SECONDARY OUTCOMES:
Change in single beat ventricular elastance | within 30 minutes after having been stabilised on the cardiothoracic ICU after performed CABG surgery
  Change in single beat ventricular elastance in reaction to both different noradrenaline doses and states of fluid responsiveness.
  Ventricular elastance (Ees) can be determined on the bedside by using a single beat measurement of left ventricular ejection fraction, stroke volume, preejection time and ejection time.
Change in single beat arterial elastance | within 30 minutes after having been stabilised on the cardiothoracic ICU after performed CABG surgery
  Change in single beat arterial elastance in reaction to both different noradrenaline doses and states of fluid responsiveness. Using an estimative formula Ea can be calculated (Ea=SBPx0.9/SV) and Ea/Ees as a marker of arterio-ventricular coupling can be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Pleym (Head of Department), md, PhD, Study Director — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Dep. for Anesthesia & Intensive care. Section of cardiothoracic Anesthesia and -intensive Care., Trondheim, Norway